CLINICAL TRIAL: NCT06648876
Title: Pharmacokinetic and Pharmacodynamics of YG1699 in Patients With Diabetes and Kidney Dysfunction
Brief Title: PK and PD of YG1699 in CKD Patients With Diabetes
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Leyi Gu, Professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-0232
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Diabetes; Renal Insufficiency, Chronic; Hemodialysis
Keywords: PK; PD; SGLT1/2 inhibitor; CKD; Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- eGFR≥30+YG1699 (Experimental): patients with eGFR ≥30ml/min/1.73M2 will be treated with YG1699 10mg QD for 8 days.
  Interventions: Drug: YG1699
- Hemodialysis+YG1699 (Experimental): patients on hemodialysis will be treated with YG1699 10mg QD for 8 days.
  Interventions: Drug: YG1699
- eGFR<20+YG1699 (Experimental): patients with eGFR <20ml/min/1.73M2 will be treated with YG1699 10mg QD for 8 days.
  Interventions: Drug: YG1699
- eGFR<20+placebo (Placebo Comparator): patients with eGFR <20ml/min/1.73M2 will be treated with placebo 10mg QD for 8 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YG1699 — 10mg qd for 8 days
  Arms: Hemodialysis+YG1699; eGFR<20+YG1699; eGFR≥30+YG1699
Drug: Placebo — 10mg qd for 8 days
  Arms: eGFR<20+placebo

SUMMARY:
The goal of this clinical trial is to learn PK and PD of YG1699 in patients with diabetes and renal dysfuction.

Participants will:

Take YG1699 or a placebo every day for 8 days. Visit the clinic 7 times for checkups and tests. Keep a diary of their symptoms. Estimate PK data from a single dose of YG1699. Estimate PD data at baseline and the last day.

DETAILED DESCRIPTION:
Background

Diabetic kidney disease (DKD), as one of the most common and serious complications of diabetes, has become the leading cause of end-stage renal disease (ESRD) worldwide. A domestic epidemiological survey shows that the prevalence of DKD in community patients was 30%-50% from 2009 to 2012, and accounted for about 40% in hospitalized patients in China. At present, the treatment of DKD is the comprehensive management of blood glucose, blood pressure and blood lipid. Nevertheless, about one-third of patients with type 1 diabetes mellitus (T1DM) and nearly half of patients with type 2 diabetes mellitus (T2DM) will progress to ESRD. Patients with DKD have higher complication rates and mortality. Studies have shown that the mortality rate of patients with diabetes complicated with DKD is 3 to 12 times higher than that of patients with simple diabetes. Although blood glucose is actively controlled and angiotensin-converting enzyme inhibitors (ACEI) or angiotensin II receptor blockers (ARB) are used to control hypertension in the treatment of diabetes, the progression of DKD is still inevitable. Much more clinical needs are still present. Sodium-glucose co-transporter inhibitors (SGLT2i) are new hypoglycemic drugs discovered in recent years. They play their hypoglycemic roles by inhibiting glucose reabsorption in renal tubules and increasing urinary glucose excretion. More clinical studies have found that SGLT2s not only the hypoglycemic effect, but also has the effect of delaying the progression of DKD and improving the prognosis of heart failure, and is recommended by international authoritative guidelines with class IA evidence for cardiorenal organ protection.

Glucose cannot freely pass through the cell membrane and must rely on glucose transporter proteins on the cell membrane. Sodium-dependent glucose cotransporters (SGLTs) are an important family of transporter proteins that regulate glucose absorption and excretion. SGLT1 and SGLT2 are the most well studied members of this family and are both major glucose transporter proteins. SGLT1 is expressed in various tissues such as the small intestine, heart and kidney. SGLT2 is mainly expressed in segment S1 of the proximal convoluted tubule of the kidney.

In the renal tubules, 95% of glucose is reabsorbed through SGLT2, and 5% of glucose is reabsorbed through SGLT1. When SGLT2 is inhibited, the glucose reabsorbed through SGLT1 significantly increases to 50%, so the hypoglycemic effect of SGLT2 inhibitors may be weakened. The dual effects of SGLT1 and SGLT2 inhibitors can bring more potential benefits for treatment, including continuing to maintain the effectiveness of SGLT2 selective inhibitors; inducing intestinal cells to secrete endogenous glucagon-like peptide-1 (GLP-1) and YY peptide (PYY); reducing the adverse reactions of SGLT2 inhibition, such as genitourinary tract infections and constipation; blocking or delaying the absorption of glucose by the gastrointestinal tract.

Sotagliflozin is a SGLT2i with partial SGLT1 inhibitory activity. It was approved by the European Medicines Agency (EMA) in 2019 for adjuvant treatment of T1DM complicated with obesity. Recently, the sotagliflozin heart failure protection study was terminated in the middle stage due to the excellent effect of improving the outcome of heart failure. And it has a good effect of reducing proteinuria in patients with DKD. This suggests that SGLT1/2 dual-channel blockers may have better hypoglycemic and organ protection effects.

YG1699 is an oral SGLT1 and SGLT2 dual-channel blocker, belonging to c-aryl glucoside derivatives. It can reduce the absorption of glucose into the blood in the gastrointestinal tract by inhibiting SGLT-1, and at the same time inhibit the reabsorption of glucose in the proximal convoluted tubule of the kidney by inhibiting SGLT-2, thereby increasing the excretion of glucose from the kidney and effectively reducing blood glucose levels. YG1699 reduces the risk of DKA caused by SGLT2i by increasing SGLT1 inhibitory activity. In addition, YG1699 shows non-pH-dependent solubility, has sufficient solubility in the gastrointestinal tract, has a high oral bioavailability in preclinical models, and has a low possibility of drug interactions. At present, including YG1699, there are three SGLT1/2 dual inhibitor are in the clinical research stage.

YG1699 has completed three clinical trials, named the phase I study (YG1699-01) on healthy subjects in the United States and the phase II study (YG1699-201) on type 1 diabetes, as well as the bridging study (YG1699-102) on healthy subjects in China. These clinical studies have confirmed that YG1699 has good human PK characteristics and good safety and tolerance. In the phase II T1DM study, compared head-to-head with DAPA, it shows a better effect on reducing postprandial blood glucose. All these clinical trials are in patients with eGFR>30 ml/min/1.73M2.

However, about 12 million diabetic patients have renal insufficiency, and there is still no pharmacokinetic and pharmacodynamic data of YG1699 in patients with renal insufficiency.

Key inclusion criteria include:

1. Ability to provide informed consent
2. Male or female patients ,age between 18 and 70 at screening
3. Meet the diagnostic criteria for diabetic nephropathy, including patients with type 1 or type 2 diabetes;
4. Fasting blood glucose <11.1 mmol/L, stable on baseline anti-diabetic medication
5. No history of SGLT2i use within the past month
6. Hemodialysis patients must have maintenance hemodialysis for more than 3 months, with 3 sessions per week (limited to HD or HDF treatment), and spKt/V>1.2 within 6 months
7. The patient has not used glucocorticoids, calcineurin inhibitors (cyclosporine, tacrolimus), etc. that affect blood sugar within the past month before signing the informed consent form
8. The baseline diabetes management medication regimen has been stable within the past 2 weeks.

Key exclusion criteria include:

1. Hypoglycemia occurs more than 2 times in one month
2. History of ketoacidosis
3. Patients who are being treated with swiram and digoxin
4. Patients with acute kidney injury (serum creatinine increased by ≥ 50% within 1 week) 5. Abnormal liver function (ALT >3 times the upper limit of normal value)

6. Hemoglobin <80g/L or >150g/L 7. The blood pressure of patients with recent symptomatic hypotension is lower than 90/60 mmHg 8. There is acute myocardial infarction stroke infection in the past month 9. There is systemic active infection or uncured tumor 10. The dialysis regimen of HD patients included HP treatment 11. Participating in other interventional clinical studies 12. Pregnant or lactating women 13. Other situations that the researcher thinks are not suitable for joining the study

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent
2. Male or female patients ,age between 18 and 70 at screening
3. Meet the diagnostic criteria for diabetic nephropathy, including patients with type 1 or type 2 diabetes;
4. Fasting blood glucose <11.1 mmol/L, stable on baseline anti-diabetic medication
5. No history of SGLT2i use within the past month
6. Hemodialysis patients must have maintenance hemodialysis for more than 3 months, with 3 sessions per week (limited to HD or HDF treatment), and spKt/V>1.2 within 6 months
7. The patient has not used glucocorticoids, calcineurin inhibitors (cyclosporine, tacrolimus), etc. that affect blood sugar within the past month before signing the informed consent form
8. The baseline diabetes management medication regimen has been stable within the past 2 weeks.

Exclusion Criteria:

1. Hypoglycemia occurs more than 2 times in one month
2. History of ketoacidosis
3. Patients who are being treated with swiram and digoxin
4. Patients with acute kidney injury (serum creatinine increased by ≥ 50% within 1 week)
5. Abnormal liver function (ALT > 3 times the upper limit of normal value)
6. Hemoglobin < 80g/L or > 150g/L
7. The blood pressure of patients with recent symptomatic hypotension is lower than 90/60 mmHg
8. There is acute myocardial infarction stroke infection in the past month
9. There is systemic active infection or uncured tumor
10. The dialysis regimen of HD patients included HP treatment
11. Participating in other interventional clinical studies
12. Pregnant or lactating women
13. Other situations that the researcher thinks are not suitable for joining the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
YG1699 concentration in plasma at different time | 0 hour (h), 0.5h, 1h, 2h, 4h, 8h and 12h after the first dose of YG1699 (Day1); 24 hours after the first dose of YG1699 (Day2 morning)
  single-dose pharmacokinetic

SECONDARY OUTCOMES:
Metabolite 1 concentration in plasma at different time | 0 hour (h), 0.5h, 1h, 2h, 4h, 8h and 12h after the first dose of YG1699 (Day1); 24 hours after the first dose of YG1699 (Day2 morning)
  single-dose pharmacokinetic
YG1699 steady-state concentration in plasma | Day 9 morning（the first day after discontinuation of the drug）
  steady-state pharmacokinetic
Metabolite 1 steady-state concentration in plasma | Day 9 morning（the first day after discontinuation of the drug）
  steady-state pharmacokinetic
Hemodialysis clearance of YG1699 | immediately before and immediately after the hemodialysis treatment on Day9
  pharmacokinetic
Hemodialysis clearance of Metabolite 1 | immediately before and immediately after the hemodialysis treatment on Day 9
  pharmacokinetic
OGTT | screen period and Day 8 (last day of medication)
  0h, 1h, 2h, 3h blood glucose after taking 75g oral glucose
24h urine glucose | screen period and Day 8 (last day of medication)

OTHER OUTCOMES:
Red blood cell count | Day9 morning（the first day after discontinuation of the drug）
White blood cell count | Day 9 morning（the first day after discontinuation of the drug）
Platelet count | Day 9 morning（the first day after discontinuation of the drug）
Hemoglobin | Day 9 morning（the first day after discontinuation of the drug）
Alanine aminotransaminase (ALT) | Day 9 morning（the first day after discontinuation of the drug）
Aspartate aminotransferase (AST) | Day 9 morning（the first day after discontinuation of the drug）
Total bilirubin | Day 9 morning（the first day after discontinuation of the drug）
Direct bilirubin | Day 9 morning（the first day after discontinuation of the drug）
Blood ketone body | Day 9 morning（the first day after discontinuation of the drug）
Blood pH | Day 9 morning（the first day after discontinuation of the drug）
Blood HCO3- concentration | Day 9 morning（the first day after discontinuation of the drug）
Serum creatinine | Day 9 morning（the first day after discontinuation of the drug）
estimated glomerular filtration rate (eGFR) | Day 9 morning（the first day after discontinuation of the drug）
Urinary albumin/creatinine ratio (UACR) | Day 9 morning（the first day after discontinuation of the drug）
ECG heart rate | Day 9 morning（the first day after discontinuation of the drug）
ECG heart rhythm | Day 9 morning（the first day after discontinuation of the drug）
ECG PR interval | Day 9 morning（the first day after discontinuation of the drug）
ECG QT interval | Day 9 morning（the first day after discontinuation of the drug）

CONTACTS AND LOCATIONS:
Overall Officials: Leyi Gu, Principal Investigator — RenJi Hospital
Locations (1):
- Department of nephrology , Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wright EM, Loo DD, Hirayama BA. Biology of human sodium glucose transporters. Physiol Rev. 2011 Apr;91(2):733-94. doi: 10.1152/physrev.00055.2009. PMID 21527736
- [Background] Powell DR, DaCosta CM, Gay J, Ding ZM, Smith M, Greer J, Doree D, Jeter-Jones S, Mseeh F, Rodriguez LA, Harris A, Buhring L, Platt KA, Vogel P, Brommage R, Shadoan MK, Sands AT, Zambrowicz B. Improved glycemic control in mice lacking Sglt1 and Sglt2. Am J Physiol Endocrinol Metab. 2013 Jan 15;304(2):E117-30. doi: 10.1152/ajpendo.00439.2012. Epub 2012 Nov 13. PMID 23149623
- [Background] Abdul-Ghani MA, DeFronzo RA. Inhibition of renal glucose reabsorption: a novel strategy for achieving glucose control in type 2 diabetes mellitus. Endocr Pract. 2008 Sep;14(6):782-90. doi: 10.4158/EP.14.6.782. PMID 18996802
- [Background] Rieg T, Masuda T, Gerasimova M, Mayoux E, Platt K, Powell DR, Thomson SC, Koepsell H, Vallon V. Increase in SGLT1-mediated transport explains renal glucose reabsorption during genetic and pharmacological SGLT2 inhibition in euglycemia. Am J Physiol Renal Physiol. 2014 Jan;306(2):F188-93. doi: 10.1152/ajprenal.00518.2013. Epub 2013 Nov 13. PMID 24226519
- [Background] Jung CH, Jang JE, Park JY. A Novel Therapeutic Agent for Type 2 Diabetes Mellitus: SGLT2 Inhibitor. Diabetes Metab J. 2014 Aug;38(4):261-73. doi: 10.4093/dmj.2014.38.4.261. PMID 25215272
- [Background] Cariou B, Charbonnel B. Sotagliflozin as a potential treatment for type 2 diabetes mellitus. Expert Opin Investig Drugs. 2015;24(12):1647-56. doi: 10.1517/13543784.2015.1100361. Epub 2015 Nov 7. PMID 26548423
- [Background] Wang Shanshan, Chen Dong, Chen Mingwei, et al. Analysis of the influence of metabolic syndrome on diabetic nephropathy in patients with type 2 diabetes [J]. Prevention and control of chronic diseases in China, 2011,19 (5):509-511.
- [Result] Levin A, Tonelli M, Bonventre J, Coresh J, Donner JA, Fogo AB, Fox CS, Gansevoort RT, Heerspink HJL, Jardine M, Kasiske B, Kottgen A, Kretzler M, Levey AS, Luyckx VA, Mehta R, Moe O, Obrador G, Pannu N, Parikh CR, Perkovic V, Pollock C, Stenvinkel P, Tuttle KR, Wheeler DC, Eckardt KU; ISN Global Kidney Health Summit participants. Global kidney health 2017 and beyond: a roadmap for closing gaps in care, research, and policy. Lancet. 2017 Oct 21;390(10105):1888-1917. doi: 10.1016/S0140-6736(17)30788-2. Epub 2017 Apr 20. PMID 28434650
- [Result] Bhatt DL, Szarek M, Steg PG, Cannon CP, Leiter LA, McGuire DK, Lewis JB, Riddle MC, Voors AA, Metra M, Lund LH, Komajda M, Testani JM, Wilcox CS, Ponikowski P, Lopes RD, Verma S, Lapuerta P, Pitt B; SOLOIST-WHF Trial Investigators. Sotagliflozin in Patients with Diabetes and Recent Worsening Heart Failure. N Engl J Med. 2021 Jan 14;384(2):117-128. doi: 10.1056/NEJMoa2030183. Epub 2020 Nov 16. PMID 33200892
- [Result] Cherney DZI, Ferrannini E, Umpierrez GE, Peters AL, Rosenstock J, Powell DR, Davies MJ, Banks P, Agarwal R. Efficacy and safety of sotagliflozin in patients with type 2 diabetes and stage 3 chronic kidney disease. Diabetes Obes Metab. 2023 Jun;25(6):1646-1657. doi: 10.1111/dom.15019. Epub 2023 Feb 28. PMID 36782093
- [Result] Shanghai Yanjian New Drug R&D Co., Ltd. Handbook for Researchers (Chinese). June 17, 2021